CLINICAL TRIAL: NCT04510441
Title: Artificial Intelligence-assisted Diagnosis and Prognostication in COVID-19 Using Electrocardiograms and Imaging
Brief Title: Artificial Intelligence-assisted Diagnosis and Prognostication in COVID-19 Using Electrocardiograms
Acronym: AI-COV-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Chelsea and Westminster NHS Foundation Trust (Other); London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20HH5967
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Coronavirus
Keywords: coronavirus; electrocardiogram; artificial intelligence; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nil intervention — Nil intervention; retrospective cohort study

SUMMARY:
Coronavirus Disease 2019 (COVID-19) has been widespread worldwide since December 2019. It is highly contagious, and severe cases can lead to acute respiratory distress or multiple organ failure. On 11 March 2020, the WHO made the assessment that COVID-19 can be characterised as a pandemic. With the development of machine learning, deep learning based artificial intelligence (AI) technology has demonstrated tremendous success in the field of medical data analysis due to its capacity of extracting rich features from imaging and complex clinical datasets. In this study, we aim to use clinical data collected as part of routine clinical care (heart tracings, X-rays and CT scans) to train artificial intelligence and machine learning algorithms, to accurately predict the course of disease in patients with Covid-19 infection, using these datasets.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) has been widespread worldwide since December 2019. It is highly contagious, and severe cases can lead to acute respiratory distress or multiple organ failure and ultimately death. The disease can be confirmed by using the reverse-transcription polymerase chain reaction (RT-PCR) test. ECGs, Chest x-rays and CT scans are rich sources of data that provide insight to disease that otherwise would not be available.

Knowing who to admit to the hospital or intensive care saves lives as it helps to mitigate resource shortages. Novel Artificial Intelligence tools such as Deep learning will allow a complex assessment of the Imaging and clinical data that could potentially help clinicians to make a faster and more accurate diagnosis, better triage patients and assess treatment response and ultimately better prediction of outcome. Our group has significant experience implementing machine learning algorithms on vast quantities of ECGs, such as from the UK Biobank, and propose to extend our techniques to data from patients with Covid-19.

This is a retrospective data study on patients with suspicious and confirmed COVID-19.

The study aims to recruit up to 2000 patients who will be referred to have ECGs, chest X-rays or CT scans at Chelsea and Westminster Hospital NHS Foundation Trust, Imperial College Healthcare NHS Trust and London North West London University Healthcare NHS Trust.

To be included in this study, the patient must:

* have ECGs, Chest x-ray and/or chest CT imaging (with or without contrast)
* laboratory Covid-19 virus nucleic acid test (RTPCR assay with throat swab samples) or clinical suspicion for Covid19 infection
* be aged >18 years Patients with suboptimal ECGs, chest radiograph and CT studies due to artefacts will be excluded. Patients will also be excluded if the time-interval between ECGs, chest CT and the RT-PCR assay was longer than 7 days.

This study received HRA and Health and Care Research Wales (HCRW) approval on 18 May 2020 following review by Research Ethics Committee at a meeting held on 13 May 2020(Protocol number: 20HH5967; REC reference: 20/HRA/2467).

ELIGIBILITY:
Inclusion Criteria:

* have ECGs, Chest x-ray and/or chest CT imaging (with or without contrast)
* positive laboratory Covid-19 virus nucleic acid test (RTPCR assay with throat swab samples) or clinical suspicion for Covid-19 infection
* be aged >18 years

Exclusion Criteria:

* Suboptimal ECGs, chest radiographs or CT studies for deep learning methods due to artefacts including severe
* motion artefacts which causes blurring of the contours of or significant artefacts due to metallic prosthesis which causes image degradation
* Time-interval between ECGs, chest CT and the RT-PCR assay was longer than 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective data study on patients with suspicious and confirmed COVID-19.
  The study aims to recruit up to 2000 patients who will be referred to have ECGs, chest X-rays or CT scans at Chelsea and Westminster Hospital NHS Foundation Trust, Imperial College Healthcare NHS Trust and London North West London University Healthcare NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of machine learning to be able to predict outcome of coronavirus (COVID-19) infection | At the end of data analyses, approximately 1 year
  Accuracy with which computer based analysis (machine learning) can diagnose and/or prognosticate Covid-19 Number of Participants With COVID19 who died or survived following hospital admission
Accuracy of machine learning to be able to predict prognosis of coronavirus (COVID-19) infection | At the end of data analyses, approximately 1 year
  Number of participants who required invasive vs non-invasive ventilation vs ward-based care vs died

SECONDARY OUTCOMES:
Accuracy of machine learning to be able to predict cardiac involvement of coronavirus (COVID-19) infection | At the end of data analyses, approximately 1 year
  Number of participants who had COVID19-related heart problems.
Accuracy of machine learning vs human assessment to diagnose coronavirus (COVID-19) infection | At the end of data analyses, approximately 1 year
  Number of participants that can be identified as having COVID19 using machine learning vs human or other clinical test or assessment

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - London North West University Healthcare NHS Trust, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Imperial College London (Hammersmith campus), London
  - St Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
This is a study using retrospective, pseudo-anonymised data that were acquired as part of routine clinical care for the patients. There are no direct risks to the patients' health. The main issues revolve around data security and storage. In order to address this, members of the direct care team who are not members of the research team will perform the pseudo-anonymisation of the data and pass a set of pseudo-anonymised data to the research team with no access to the pseudo-anonymisation code. The research team will therefore be unable to identify the patients from those data. The pseudo-anonymised data will also be securely stored to further minimise risks.
Supporting Information: Study Protocol, SAP
Time Frame: within study duration
Access Criteria: Researchers of the study

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT04510441/Prot_SAP_000.pdf